CLINICAL TRIAL: NCT04394052
Title: Novel Imaging Techniques for the Characterization of Musculoskeletal Tumors II: Texture Analysis and Artificial Intelligence
Brief Title: Novel Imaging Techniques for the Characterization of Musculoskeletal Tumors II
Acronym: TUMOSTEO II
Status: Recruiting | Type: Observational
Sponsor: Central Hospital, Nancy, France (Other)
Collaborators: Lorraine Cancer Institute - ICL (Unknown); Emille Gallé Surgical Center - CCEG (Unknown); Diagnostic and Interventional Adaptative Imaging Laboratory - IADI (Unknown)
Responsible Party: Sponsor
Other Study IDs: 2019PI253
Record Dates: First submitted 2020-05-12; First posted 2020-05-19 (Actual); Last update posted 2020-07-21 (Actual); Status verified 2020-05

CONDITIONS: Soft Tissue Neoplasm; Bone Neoplasm
Keywords: MRI; CT; Texture analysis; Ultra-high resolution; Tumors; Musculoskeletal
MeSH Terms: conditions — Soft Tissue Neoplasms; Bone Neoplasms; Neoplasms | interventions — Magnetic Resonance Imaging

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Soft-tissue tumors: Benign and malignant soft tissue masses
  Interventions: Diagnostic Test: MR imaging
- Bone tumors: Benign and malignant bone focal bone lesions
  Interventions: Diagnostic Test: MR imaging

INTERVENTIONS:
Diagnostic Test: MR imaging — Medical imaging
  Other Names: Ultra-high resolution CT

SUMMARY:
This study aims at evaluating the value of various artificial intelligence based techniques to improve the characterization and image post-processing for patients with musculoskeletal tumors.

DETAILED DESCRIPTION:
Comparison of values relating to the texture parameters of tumors evaluated by MRI and ultra-high resolution CT between benign and malignant lesions using histological analysis as the standard of reference.

Comparison of the diagnostic performance of texture parameters derived from different MRI sequences and ultra-high resolution CT for musculoskeletal tumor characterization.

Evaluate the impact of ultra-high resolution with respect to standard resolution on CT images Comparison of the diagnostic performance of the texture parameters for the tumor on the diagnostic performance of texture analysis derived parameters for the characterization of musculoskeletal tumors.

Evaluate the effectiveness and accuracy of automatic artificial intelligence (AI) based tumor segmentation tools.

Evaluate the use of trabecular analysis on ultra-high resolution CT images for the evaluation of tumor-bone interfaces.

ELIGIBILITY:
Inclusion Criteria:

* Patients suspected to have a bone or soft-tissue tumor referred for imaging for initial tumors characterization and staging.

Exclusion Criteria:

* Pregnancy
* Breast feeding patients
* Renal insufficiency
* Contra indications to MRI or CT
* Prior surgery or treatment to the evaluated lesion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with soft-tissue and bone tumors evaluated with MR and ultra-high resolution CT.
Sampling Method: Non-Probability Sample
Enrollment: 740 (Estimated)
Dates: Start 2020-06-01 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2030-06-01 (Estimated)

PRIMARY OUTCOMES:
Lesion benignancy or malignancy | Performed up to 6 months after CT and Magnetic Resonance (MR) imaging
  Histologic determination of lesion aggressiveness (benign versus malignant) on core biopsy material

SECONDARY OUTCOMES:
Sarcoma FNCLCC (fédération Nationale des Centres de Lutte Contre le Cancer) grade | Performed up to 1 year after CT and MR imaging
  Histologic grade of the sarcomas included in the study population with surgical resection material

CONTACTS AND LOCATIONS:
Locations (1):
- CHU-Nancy, Nancy, Lorraine, France

IPD SHARING:
Plan to Share IPD: No